CLINICAL TRIAL: NCT02843568
Title: Improving Pulmonary Function Following Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW16037; NCI-2016-01085 (Registry Identifier: NCI Trial ID); 2016-0610 (Other: Institutional Review Board); A539933 (Other: UW Madison); SMPH\VOLUNTEER STAFF\HUM ONCOL (Other: UW Madison); Protocol Version 6/9/2022 (Other: UW Madison); R01CA166703 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (Active Comparator): Subjects undergo four-dimensional computed tomographic imaging (4DCT) scans: 1 at simulation, and 2 scans at each of the 3 post-radiation therapy time points (3, 6, and 12 months). 4DCT determines lung tissue elasticity and for standard of care radiation treatment planning. Subjects undergo laboratory biomarker analysis, including spirometry, diffusion capacity (DLCO), and lung volumes (FEV, FEV1). Subjects complete a self-assessment, RTOG defined acute evaluation toxicity evaluation, RTOG late toxicity evaluation, and constitutional assessment.
  Radiation doses between 60-66 Gy using standard fractionation (1.8-2.0 Gy/fx) and 40-60 Gy stereotactic body radiation therapy (SBRT) hypofractionation schemes are utilized. Treatment volumes are at the discretion of the treating radiation oncologist and should follow standard of care.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Standard fractionation; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Four Dimensional Computed Tomographic Imaging (4DCT)
- Pulmonary Function Damage Reduction (Experimental): All criteria and specifications in the standard of care arm are applicable for this arm, including the same 4DCT scans, and laboratory biomarker analysis. Subjects randomized to this arm of the trial will have the same prescribed radiation dose to the tumor volume and held to the same radiation dose criteria as the subjects in the standard of care arm (60-66 Gy using standard fractionation (1.8-2.0 Gy/fx) and 40-60 Gy stereotactic body radiation therapy (SBRT) hypofractionation). The fundamental difference will be radiation doses for these subjects will be redistributed away from regions predicted to cause the greatest reduction in pulmonary function if damaged.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Standard fractionation; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Four Dimensional Computed Tomographic Imaging (4DCT)

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Standard fractionation — 60-66y Gy delivered in 1.8-2.0 Gy fractions over 30-36 treatments
  Other Names: Cancer Radiotherapy; Radiation
Radiation: Stereotactic Body Radiation Therapy (SBRT) — 40-60 Gy delivered in 5-20 Gy fractions over 3-8 treatments
  Other Names: SBRT; Cancer Radiotherapy; Radiation
Procedure: Four Dimensional Computed Tomographic Imaging (4DCT) — Subjects undergo a total of 7 research-ordered four dimensional computed tomographic imaging (4DCT) scans: 1 at simulation, and 2 scans at each of the 3 post-radiation therapy time points (3, 6, and 12 months). 4DCT determines lung tissue elasticity and for standard of care radiation treatment planning.
  Other Names: 4DCT

SUMMARY:
The purpose of this study is to develop radiation plans that will help preserve lung function in healthy tissue surrounding the tumor. We believe that 4DCT scans can be useful in designing radiation treatment plans that help us avoid healthy normal functioning lung tissue close to lung tumors. Currently 4DCT scans are used to help us determine exactly where the tumor is and how it moves when you breathe. In this study we will also use the 4DCT scans to try to identify high functioning normal lung tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of non-small cell lung cancer or lung metastasis from a solid tumor. One biopsy site is adequate for multiple sites of thoracic disease.
* Treatment includes localized radiation therapy with or without chemotherapy
* Karnofsky ≥ 60%
* Not pregnant per radiation oncology standard procedures
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior (within last 6 months) or future planned therapeutic surgery for the treatment of the existing lung cancer
* Prior thoracic radiotherapy
* Severe COPD defined as disease requiring an inpatient stay for respiratory deterioration within the past 3 months
* Oxygen dependence of > 2 L/min continuously throughout the day at baseline
* Known underlying collagen vascular disease or intrinsic lung disease that could complicate expected sequelae of radiation (idiopathic pulmonary fibrosis, Wegener's granulomatosis)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carri K Glide-Hurst, PhD, DABR, FAAPM, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Baschnagel AM, Flakus MJ, Wallat EM, Wuschner AE, Chappell RJ, Bayliss RA, Kimple RJ, Christensen GE, Reinhardt JM, Bassetti MF, Bayouth JE. A Phase 2 Randomized Clinical Trial Evaluating 4-Dimensional Computed Tomography Ventilation-Based Functional Lung Avoidance Radiation Therapy for Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2024 Aug 1;119(5):1393-1402. doi: 10.1016/j.ijrobp.2024.02.019. Epub 2024 Feb 20. PMID 38387810
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Subjects undergo four-dimensional computed tomographic imaging (4DCT) scans: 1 at simulation, and 2 scans at each of the 3 post-radiation therapy time points (3, 6, and 12 months). 4DCT determines lung tissue elasticity and for standard of care radiation treatment planning. Subjects undergo laboratory biomarker analysis, including spirometry, diffusion capacity (DLCO), and lung volumes (FEV, FEV1). Subjects complete a self-assessment, RTOG defined acute evaluation toxicity evaluation, RTOG late toxicity evaluation, and constitutional assessment.
  Radiation doses between 60-66 Gy using standard fractionation (1.8-2.0 Gy/fx) and 40-60 Gy stereotactic body radiation therapy (SBRT) hypofractionation schemes are utilized. Treatment volumes are at the discretion of the treating radiation oncologist and should follow standard of care.
  Laboratory Biomarker Analysis: Correlative studies
  Standard fractionation: 60-66y Gy delivered in 1.8-2.0 Gy fractions over 30-36 treatments
  Stereotactic Body Radiation Therapy (SBRT): 40-60 Gy delivered in 5-20 Gy fractions over 3-8 treatments
  Four Dimensional Computed Tomographic Imaging (4DCT): Subjects undergo a total of 7 research-ordered four dimensional computed tomographic imaging (4DCT) scans: 1 at simulation, and 2 scans at each of the 3 post-radiation therapy time points (3, 6, and 12 months). 4DCT determines lung tissue elasticity and for standard of care radiation treatment planning.
Period: Overall Study
Arm/Group | Standard of Care | Pulmonary Function Damage Reduction
Started | 65 | 57
Evaluable for Primary Analysis (Participants were excluded as they had a change in treatment.) | 61 | 55
SBRT Cohort (Analyzed for Toxicities) | 30 | 31
Conventional Cohort (Analyzed for Toxicities) | 31 | 24
Participants at 3 Months | 57 | 51
Participants at 6 Months | 53 | 43
Participants at 12 Months | 43 | 34
Analyzed for Primary Endpoints | 55 | 51
Completed | 55 | 51
Not Completed | 10 | 6
Not completed — Excluded from Primary Population due to change in treatment | 4 | 2
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable for Primary Analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Pulmonary Function Damage Reduction | Total
Number analyzed (Participants) | 61 | 55 | 116
Age, Customized [Median (Full Range); unit: years]
  median age | 69 [49 to 89] | 71 [52 to 88] | 70 [49 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 32 | 56
  Male | 37 | 23 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 61 | 55 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 58 | 53 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 55 | 116

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function, Based on Changes in Tissue Elasticity Measured From 4DCT
Description: The primary endpoint of this study will be the ratio of the tissue elasticity map following RT to the elasticity map before RT (i.e., the Jacobian ratio of (post RT /pre RT)) calculated from 4DCT at 3 months post-RT. Based on the randomness of our measurement technique, diminished expansion (i.e. substantial change) is defined as a Jacobian ratio <0.94 (i.e., less than 94% of the pre-RT value).
Time Frame: 3 months post RT
Measure: Median (Full Range); unit: ratio
Arm/Group | Standard of Care | Pulmonary Function Damage Reduction
Number analyzed (Participants) | 55 | 51
ratio | 1.09 [0.42 to 2.8] | 1.13 [0.37 to 3.2]

2. Secondary Outcome: Temporal Changes in Reduced Elasticity Determined by the Volume of Lung Where Expansion is Improved
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: During therapy to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

3. Secondary Outcome: Temporal Changes in Increased Elasticity Determined by the Volume of Lung Where Expansion is Improved
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: During therapy to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

4. Secondary Outcome: Temporal Changes in Fraction of Expanding Lung Determined by the Volume of Lung Where "Meaningful" Expansion Occurs
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: During therapy to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

5. Secondary Outcome: Validation in Consistency of Tissue Elasticity Changes Measured With Values Predicted Based on Existing Radiation Dose Response Curves
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: Up to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

6. Secondary Outcome: Median Absolute Change in the Percent Predicted for Pulmonary Function Tests (PFTs)
Description: Median absolute change in the percent predicted following pulmonary function tests reported: Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), and diffusing capacity of carbon monoxide (DLCO). All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: Pre-RT up to 12 months post-RT
Population: This measures a change from baseline, not all participants completed all time points
Measure: Median (Full Range); unit: percent predicted
Groups:
- Standard of Care: Conventionally Fractionated Cohort; Pulmonary Function Damage Reduction: Conventionally Fractionated Cohort: Standard fractionation: 60-66y Gy delivered in 1.8-2.0 Gy fractions over 30-36 treatments
- Standard of Care: SBRT Cohort: Participants undergoing stereotactic body radiation therapy (SBRT) 40-60 Gy delivered in 5-20 Gy fractions over 3-8 treatments
- Pulmonary Function Damage Reduction: SBRT Cohort: Participants undergoing Stereotactic Body Radiation Therapy (SBRT): 40-60 Gy delivered in 5-20 Gy fractions over 3-8 treatments
Arm/Group | Standard of Care: Conventionally Fractionated Cohort | Pulmonary Function Damage Reduction: Conventionally Fractionated Cohort | Standard of Care: SBRT Cohort | Pulmonary Function Damage Reduction: SBRT Cohort
Number analyzed (Participants) | 31 | 23 | 30 | 30
percent predicted
  Median Absolute Change in the FEV1 percent predicted from baseline to 3 months: number analyzed (Participants) | 27 | 22 | 29 | 29
  Median Absolute Change in the FEV1 percent predicted from baseline to 3 months | -5 [-28 to 10] | -3 [-12 to 46] | -2 [-15 to 10] | -2 [-21 to 18]
  Median Absolute Change in the FEV1 percent predicted from baseline to 6 months: number analyzed (Participants) | 24 | 15 | 29 | 27
  Median Absolute Change in the FEV1 percent predicted from baseline to 6 months | -4 [-32 to 14] | -4 [-15 to 13] | -2 [-31 to 13] | -3 [-24 to 19]
  Median Absolute Change in the FEV1 percent predicted from baseline to 12 months: number analyzed (Participants) | 15 | 11 | 25 | 23
  Median Absolute Change in the FEV1 percent predicted from baseline to 12 months | 2 [-26 to 23] | 12 [-36 to 25] | -2 [-18 to 12] | -1 [-29 to 18]
  Median Absolute Change in the FVC percent predicted from baseline to 3 months: number analyzed (Participants) | 27 | 22 | 29 | 29
  Median Absolute Change in the FVC percent predicted from baseline to 3 months | -6 [-34 to 11] | 1.5 [-15 to 28] | 0 [-15 to 30] | 0 [-20 to 24]
  Median Absolute Change in the FVC percent predicted from baseline to 6 months: number analyzed (Participants) | 24 | 15 | 29 | 27
  Median Absolute Change in the FVC percent predicted from baseline to 6 months | -4.5 [-35 to 20] | -2 [-21 to 27] | -0.5 [-41 to 30] | -2 [-18 to 20]
  Median Absolute Change in the FVC percent predicted from baseline to 12 months: number analyzed (Participants) | 15 | 11 | 25 | 23
  Median Absolute Change in the FVC percent predicted from baseline to 12 months | -5 [-20 to 29] | 8 [-36 to 21] | 0 [-19 to 15] | 2 [-26 to 27]
  Median Absolute Change in the DLCO percent predicted from baseline to 3 months: number analyzed (Participants) | 27 | 22 | 29 | 29
  Median Absolute Change in the DLCO percent predicted from baseline to 3 months | -12 [-57 to 12] | -11 [-29 to 4] | -2.5 [-21 to 33] | -2 [-52 to 22]
  Median Absolute Change in the DLCO percent predicted from baseline to 6 months: number analyzed (Participants) | 24 | 15 | 29 | 27
  Median Absolute Change in the DLCO percent predicted from baseline to 6 months | -11 [-62 to 15] | -9.5 [-33 to 7] | -6.5 [-31 to 15] | -0.5 [-43 to 24]
  Median Absolute Change in the DLCO percent predicted from baseline to 12 months: number analyzed (Participants) | 15 | 11 | 25 | 23
  Median Absolute Change in the DLCO percent predicted from baseline to 12 months | 12 [-24 to 48] | 5 [-9 to 43] | 2.5 [-37 to 48] | 1 [-36 to 55]

7. Secondary Outcome: Change in Level of Plasma TGF-beta
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: Baseline up to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

8. Secondary Outcome: Change in Level of Plasma Cytokines
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: Baseline up to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

9. Secondary Outcome: Variation of the Tissue Elasticity Calculated Between Scan 1 and Scan 2 at Each Time Point Will be Quantified and Compared to Longitudinal Changes in Tissue Elasticity
Description: All statistical tests will be two-sided and assessed for significance at the 5% level.
Time Frame: Up to 12 months post-RT
Reporting Status: Not Posted, anticipated posting 2025-04

ADVERSE EVENTS:
Time Frame: SAEs were collected for 3 months, Other Adverse Events were collected for 12 months, All Cause mortality was collected for 30 days post-RT
Arm/Group | Standard of Care | Pulmonary Function Damage Reduction
All-Cause Mortality (participants affected / at risk) | 3/61 | 3/55
Serious Adverse Events (participants affected / at risk) | 7/61 | 10/55
Other Adverse Events (participants affected / at risk) | 61/61 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=61) | Pulmonary Function Damage Reduction (N=55)
Death NOS (General disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=61) | Pulmonary Function Damage Reduction (N=55)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Esophagitis (Gastrointestinal disorders) | 15 | 10
Rib fracture (General disorders) | 4 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Other- FEV (Respiratory, thoracic and mediastinal disorders) | 23 | 17
Other - DLCO (Respiratory, thoracic and mediastinal disorders) | 38 | 28
SVT arrhythmia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02843568/Prot_SAP_000.pdf